CLINICAL TRIAL: NCT01738438
Title: A Phase II Study of XL184 (Cabozantinib) for Metastatic Triple-Negative Breast Cancer
Brief Title: Cabozantinib for Metastatic Triple Negative BrCa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Sara Tolaney, Prinicipal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-431
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Results first posted 2016-07-07 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
Keywords: Metastatic; Triple Negative; Stage IV
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabozantinib (Experimental): Cabozantinib was given at a dose of 60 mg orally once per day for 21 day cycles. Treatment continued in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib
  Other Names: XL184

SUMMARY:
In this research study, we are looking at the anti-tumor effects of Cabozantinib (XL184) in metastatic breast cancer. Data suggest that MET expression and activation are important for initiation and progression of triple-negative breast cancer (TNBC). We evaluated the efficacy of cabozantinib (XL184), a novel inhibitor of multiple receptor tyrosine kinases, including MET and VEGFR2, in patients with metastatic TNBC.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the activity of cabozantinib, as defined by objective response rate in patients with triple-negative metastatic breast cancer

Secondary

* To evaluate progression free survival
* To evaluate c-Met and phospho c-Met expression in archival tumor tissue
* To evaluate the incidence of c-Met amplified circulating tumor cells at baseline
* To evaluate potential plasma biomarkers of cabozantinib

DESIGN:

This study uses a two-stage design enrolling 35 patients to evaluate efficacy of cabozantinib based on overall response defined as complete or partial response per RECIST1.1 criteria. The null and alternative overall response rates were 5% and 20%. If one or more patients enrolled in the stage one cohort (n=13 patients) achieve PR or better then accrual proceeds to stage two (n=22 patients).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast cancer with stage IV disease
* Primary tumor and/or metastasis must be ER-negative, PR-negative and HER2-negative
* May have received 0-3 prior chemotherapeutic regimens for metastatic breast cancer. Must be off treatment for at least 21 days prior to enrollment
* Must have discontinued all biologic therapy at least 14 days before enrollment
* May have received prior radiation therapy in the early stage or metastatic setting, but must have completed treatment at least 14 days prior to enrollment
* Must agree to use medically acceptable methods of contraception
* Confirmed availability of formalin-fixed, paraffin-embedded tumor tissue
* Able to swallow tablets

Exclusion Criteria:

* Pregnant or breastfeeding
* Received another investigational agent within 14 days prior to enrollment
* Received prior c-Met inhibitor
* Known brain metastases that are untreated, symptomatic or require therapy to control symptoms
* Psychiatric illness or social situation that could limit ability to comply with study requirements
* Require concomitant treatment in therapeutic doses with anticoagulants or antiplatelet agents
* Diagnosis of another malignancy requiring systemic treatment within the last two years (except non-melanoma skin cancer or in-situ carcinoma of the cervix)
* Known to be positive for HIV
* Active infection requiring IV antibiotics at Day 1 of cycle 1
* Uncontrolled, significant intercurrent illness
* Requires chronic concomitant treatment of a strong CYP3A4 inducer
* tumor in contact with, invading or encasing major blood vessels
* Have experienced clinically significant gastrointestinal bleeding within 6 months, hemoptysis of more than 0.5 teaspoon of red blood within 3 months or other signs indicative of pulmonary hemorrhage within 3 months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute at Faulkner Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weber ZT, Collier KA, Tallman D, Forman J, Shukla S, Asad S, Rhoades J, Freeman S, Parsons HA, Williams NO, Barroso-Sousa R, Stover EH, Mahdi H, Cibulskis C, Lennon NJ, Ha G, Adalsteinsson VA, Tolaney SM, Stover DG. Modeling clonal structure over narrow time frames via circulating tumor DNA in metastatic breast cancer. Genome Med. 2021 May 20;13(1):89. doi: 10.1186/s13073-021-00895-x. PMID 34016182

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from January 2013 through June 2014.
Period: Overall Study
Arm/Group | Cabozantinib
Started | 35
Completed | 0 (Since treatment was not of fixed duration, all participants were considered as 'Not Completed'.)
Not Completed | 35
Not completed — Disease Progression | 32
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all treated patients.
Arm/Group | Cabozantinib
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 50 [31 to 78]
Gender [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The objective response rate (ORR) was defined as achieving complete response (CR) or partial response (PR) on treatment based on RECIST1.1 criteria. For target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions. Confirmatory scans were required 3 weeks following initial documentation.
Time Frame: Disease was evaluated radiologically at baseline, week 6 and every 9 weeks on treatment; Treatment continued until disease progression or unacceptable toxicity. Treatment duration was a median of 3 cycles range (1-17).
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 35
proportion of participants | 0.09 [0.02 to 0.26]

2. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) estimated using Kaplan-Meier methods was defined as the time from registration to documented disease progression (PD) or death. Based on RECIST1.1, radiographic PD is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum since beginning therapy, the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Patients who were event-free were censored at the date of their last disease evaluation.
Time Frame: as for outcome 1
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib
Number analyzed (Participants) | 35
months | 2 [1.3 to 3.3]

3. Post Hoc Outcome: 15-Week Clinical Benefit Rate
Description: The 15-week clinical benefit rate (CBR) was defined as absence of disease progression (PD) per RECIST1.1 criteria at the second disease assessment (week 15). Radiographic PD is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum since beginning therapy, the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Confirmatory scans for response were required 3 weeks following initial documentation.
Time Frame: Disease was evaluated radiologically at baseline, week 6 and week 15 on treatment.
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 35
proportion of participants | .34 [.19 to 0.52]

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment. Treatment duration in cycles was a median (range) of 3 (1-17).
Description: Maximum grade toxicity by type for a patient over time including only events with possible, probable or definite attribution was first calculated. Patients appear once for a given toxicity type. Serious and Other AEs were defined as events of grades 3-5 and grades1-2, respectively, based on CTCAEv3. 'Other' events have no further specification.
Arm/Group | Cabozantinib
Serious Adverse Events (participants affected / at risk) | 14/35
Other Adverse Events (participants affected / at risk) | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=35)
Infections and infestations - Other (Infections and infestations) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Lipase increased (Investigations) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=35)
Anemia (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 6
Eyelid function disorder (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 14
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 10
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 19
Fatigue (General disorders) | 26
Malaise (General disorders) | 2
Mucosal infection (Infections and infestations) | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 3
Serum amylase increased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Investigations - Other (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 12
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 3
Dysgeusia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Psychiatric disorders - Other (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Irregular menstruation (Reproductive system and breast disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1
Nail loss (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 7
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes